CLINICAL TRIAL: NCT05138666
Title: Non-invasive Tools to Better Diagnose Invasive Aspergillosis Infections in ICU Patients With COVID-19 and Other Non-immunosuppressive Conditions.
Brief Title: Non-invasive Tools to Diagnose Invasive Aspergillosis Infections in ICU Patients With COVID-19 and Other Conditions.
Acronym: BM-ASP-ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/656
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Invasive Pulmonary Aspergillosis
Keywords: ICU patients; Covid-19
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biological sample (Experimental): respiratory and blood sample
  Interventions: Biological: respiratory sample; Biological: blood sample

INTERVENTIONS:
Biological: respiratory sample — tracheal aspirate or sputum if the patient is not intubated
Biological: blood sample — Blood sampling drawn from an existing arterial line twice a week

SUMMARY:
Invasive aspergillosis (IA) are difficult to diagnose in the ICU population, as the patients often do not present the conventional risks factors of immunocompromised patients (EORTC/MSG criteria). In the ICU population, patients often present other risk factors, such as cirrhosis, COPD, influenza and currently SARS-Cov2. The clinicians are thus currently missing precise criteria to distinguish colonization from IA in these patients, while they need to decide if an antifungal treatment is necessary or not.

A new algorithm, entitled BM ASP ICU, based on investigators field experience and the scientific literature, which takes into account both EORTC/MSG criteria and a combination of fungal biomarkers, was proposed recently by Haman et al, Annals Intensive Care, 2021. Additional serological assays (immunoprecipitation and ELISA) showed since their interest, especially concerning SARS-Cov2 patients, a new population at risk of IA in the ICU, which emerged in the past months.

The present study aims at prospectively implementing the BM ASP ICU algorithm during two years in the routine practice of six ICU units distributed in general and teaching hospitals situated northeast of France. The BM ASP ICU algorithm would be completed by serological assays aiming at assessing a sensitization towards Aspergillus fumigatus.

The investigators plan to include 400 ICU patients at risk of IA; SARS-Cov2 patients will be part of the cohort. A weekly screening including culture of respiratory samples, galactomannan antigen, fungal qPCRS (targeting A. fumigatus), and A. fumigatus serology will be applied for all included patients.

The performance (sensitivity and specificity, likelihood ratios) of each fungal biomarkers, alone and in combination with others, will be assessed, for all patients, and also within subgroups of patients with specific risk factors (such as SARS-Cov2 for example).

These results should lead to solid understanding of which combination of tests is optimal to diagnose IA and thus to initiate appropriate antifungal treatment. the investigators hope that this study will result in improved survival rate of ICU patients with IA.

ELIGIBILITY:
Inclusion Criteria:

1. ICU adult patient (age > 18 years old at inclusion)
2. Patient with respiratory distress (fever refractory to > 3 days of antibiotherapy, pleuritic chest pain, hemoptysis) or Patient with sign of infection on thoracic scan or Patient with positive culture for Aspergillus sp on any respiratory sample
3. Informed consent signed by the patient or proxy
4. Patient with health insurance

Exclusion Criteria:

1. Minor patient (age < 18 years old at inclusion)
2. Known risk of immunodepression as defined by EORTC/MSG:

   * Recent history neutropenia (< 500 neutrophils/mm3 for > 10 days)
   * Haematological malignancy
   * Receipt of an allogenic stem cell transplant
   * Receipt of a solid organ transplant
   * Prolonged use of corticosteroids (excluding among patients with allergic bronchopulmonary aspergillosis) at a therapeutic dose of ≥0·3 mg/kg corticosteroids for ≥3 weeks in the past 60 days
   * Treatment with recognized T-cell immunosuppressant for more than 90 days (such as calcineurin inhibitors, TNF blockers, lymphocyte-specific monoclonal antibodies, and immunosuppressive nucleoside analogues)
   * Treatment with recognized inhibitors of B-cell receptor pathway (e. g, ibrutinib), possibly BCL2 inhibitors (e. g, venetoclax)
   * Inherited severe immunodeficiency (e. g, chronic granulomatous disease, STAT3 deficiency, or severe combined immunodeficiency)
   * Acute graft-versus-host disease grade III or IV, involving the gut, lungs, or liver, that is refractory to first-line treatment with steroids
3. Patient under legal protection (e. g, tutorship)
4. Patients without health insurance
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Performance indicators of the algorithm | 90 days
  sensitivity, specificity, positive and negative predictive values, and likelihood ratios.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Chrisptophe NAVELLOU, MD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No